CLINICAL TRIAL: NCT02352272
Title: Benefits of Sleep Extension on Cognitive and Physical Performances During Baseline, Total Sleep Deprivation and Recovery (BankingSleep)
Brief Title: Benefits of Sleep Extension on Performances During Total Sleep Deprivation (BankingSleep)
Acronym: BankingSleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Principal Investigator, Fabien SAUVET, Docteur, Institut de Recherche Biomedicale des Armees
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14ca703op1; 2013-A01403-42 (Other: ANSM ID RCB)
Record Dates: First submitted 2015-01-19; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Sleep Deprivation
Keywords: sleep extension; attention; physical performance
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep extension (Experimental): Subject spend 10 hours Time in bed per day during 6 nights. This period is follow by a total sleep deprivation intervention (i.e. 39 hours awaking) in laboratory.
  Interventions: Other: Total Sleep deprivation
- Habitual sleep (Sham Comparator): Subject respect their habitual Time in bed during 6 nights. This period is follow by a total sleep deprivation intervention (i.e. 39 hours awaking) in laboratory.
  Interventions: Other: Total Sleep deprivation

INTERVENTIONS:
Other: Total Sleep deprivation — Subject are submitted to 39 hours of continuous awaking in laboratory and a recovery night
  Other Names: TSD

SUMMARY:
Objectives: investigate the effects of 6 nights of sleep extension on physical and cognitive performances before, during total sleep deprivation (39 hours continuous awaking) and after a subsequent recovery sleep.

Design: Subjects participated in two experimental conditions (randomized cross-over design): extended sleep (10-h in bed, EXT) and habitual sleep (8-h in bed, HAB). In each condition, subjects performed two consecutive phases: (1) six nights of either EXT or HAB (2) three experiments days in-laboratory:baseline (BASE), sleep deprivation (TSD) and after 10 h of recovery sleep(REC). Performance tests were administered every 3 hours over the 3-d in laboratory.

Setting: This cross-over and randomized study was conducted under standardized laboratory conditions with continuous polysomnographic recording Participants: 14 healthy men (age range: 26-37 years) participated in the study.

Interventions: EXT vs. HAB sleep durations prior to total sleep deprivation (39 hr continuous awaking).

DETAILED DESCRIPTION:
Many human endeavors require high-level cognitive performance situations (e.g., health care, military operations, space flight) along the whole nycthemera (i.e. the 24-h cycle).

It has long been established that both acute total sleep deprivation (TSD) and chronic sleep restriction impair ability to maintain wakefulness, increase subjective sleepiness and sleep propensity, and most critically reduce various aspects of cognitive performance. In studies conducted in both laboratory setting and different professional situations inducing insufficient sleep, the most consistently and dramatically impacted cognitive capacities were sustained attention and alertness. This degradation of cognitive performance after a period of sleep deprivation is linked to an increase of sleep pressure, e.g. a reduction in the latency to sleep onset or increase of number of involuntary micro sleeps.

To identify countermeasures to deleterious effects of sleep deprivation is critical in many professional areas.

Management of wake/sleep cycle appears to have an important impact of alertness during sleep deprivation (e.g. sleep habits or physical activity, see the review. Recently, Rupp and coll. (2012) reported that one week of sleep extension realized before one week of sleep restriction (3 h/night) influence the rate of degradation of cognitive performance and alertness during this period and the subsequent recovery period. In other words, they proposed that sleep can be "banked" before a period of sleep loss and may help sustain performance and alertness. With a different experimental paradigm (i.e. without subsequent sleep deprivation), studies have shown that sleep extension (realized over different periods of time) may improve physical performance, attentional performance, or mood. The fact of increasing total sleep time over a period of time represents an attractive non-pharmacological countermeasure to limit the deleterious effects on performance induced by sleep privation. However, there is no study with cross-over and randomized design to assess effect on relatively short period (6 nights) of sleep extension on performance before, during total sleep deprivation and recovery. Moreover, there is no direct measurement of sleep pressure as continuous EEG monitoring to quantify micro sleep episode during period of sleep deprivation and effect of sleep extension on physical performance is not known.

Hence, the aim of this study was to assess the effects of 6 nights of sleep extension (EXT) on physical and cognitive performances, alertness and homeostatic sleep pressure before, during total sleep deprivation and the subsequent recovery day.

The investigators hypothesized that EXT would: i) partly prevents the physical and cognitive performances degradation-induced by total sleep deprivation ii) decreases the sleep pressure before, during and after total sleep deprivation and iii) improves the recovery speed of physical and cognitive performances.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject
* voluntary

Exclusion Criteria:

* an average of > 9 h and < 6 h sleep per night
* a difference > 45 min between week night and weekend night
* sleep debt
* sleep disorders
* medication
* alcool or toxic consumption
* up to 300 mg caffeine per day consumption
* neurologic, cardiovascular, metabolic, pulmonary psychiatric disease or disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of errors during PVT (n) | Every 3 hours, up to 24 hours of baseline, total sleep deprivation (TSD), and recovery
  number of errors (<100ms or > 500ms) during a10 min Psychomotor Vigilance test (PVT)

SECONDARY OUTCOMES:
median speed during PVT (s-1) | Every 3 hours, up to 24 hours of baseline, total sleep deprivation (TSD), and recovery
  median speed response during a10 min Psychomotor Vigilance test (PVT)
number of micro sleep (n) | Every 3 hours, up to 24 hours of baseline, total sleep deprivation (TSD), and recovery
  number of micro sleep (> 5 sec) per hour during baseline, TSD and recovery
Sleep latency (min) | Every 3 hours, up to 24 hours of baseline, total sleep deprivation (TSD), and recovery
  Sleep latency during multiple sleep latency test (MSLT)
Muscular force (dyn) | At 10:00 on D1 (Baseline), D2 (TSD) and D3 (Recovery)
  Muscular force developed by the subject
Response to Trans Magnetic Stimulation (%) | At 10:00 on D1 (Baseline), D2 (TSD) and D3 (Recovery)
  Effect of trans magnetic stimulation on Muscular force developed by the subject
Polysomnographic classification (N1, N2, N3, REM) | night during DA (Baseline) and D3 (Recovery)
  Evaluation of the duration of each sleep stages during the night before and after TSD

CONTACTS AND LOCATIONS:
Overall Officials: Damien LEGER, MD, PhD, Study Chair — Sleep center, Hotel Dieu Paris; Mounir CHENNAOUI, PhD, Study Director — Institut de Recherche Biomedicale des Armees; Fabien SAUVET, MD, PhD, Principal Investigator — Institut de Recherche Biomedicale des Armees
Locations (1):
- Hotel Dieu Hospital, Paris, France

REFERENCES:
- [Background] Rupp TL, Wesensten NJ, Bliese PD, Balkin TJ. Banking sleep: realization of benefits during subsequent sleep restriction and recovery. Sleep. 2009 Mar;32(3):311-21. doi: 10.1093/sleep/32.3.311. PMID 19294951
- [Background] Chennaoui M, Sauvet F, Drogou C, Van Beers P, Langrume C, Guillard M, Gourby B, Bourrilhon C, Florence G, Gomez-Merino D. Effect of one night of sleep loss on changes in tumor necrosis factor alpha (TNF-alpha) levels in healthy men. Cytokine. 2011 Nov;56(2):318-24. doi: 10.1016/j.cyto.2011.06.002. Epub 2011 Jul 6. PMID 21737301
- [Background] Sauvet F, Leftheriotis G, Gomez-Merino D, Langrume C, Drogou C, Van Beers P, Bourrilhon C, Florence G, Chennaoui M. Effect of acute sleep deprivation on vascular function in healthy subjects. J Appl Physiol (1985). 2010 Jan;108(1):68-75. doi: 10.1152/japplphysiol.00851.2009. Epub 2009 Nov 12. PMID 19910332
- [Background] Chennaoui M, Arnal PJ, Sauvet F, Leger D. Sleep and exercise: a reciprocal issue? Sleep Med Rev. 2015 Apr;20:59-72. doi: 10.1016/j.smrv.2014.06.008. Epub 2014 Jun 30. PMID 25127157
- [Background] Temesi J, Arnal PJ, Davranche K, Bonnefoy R, Levy P, Verges S, Millet GY. Does central fatigue explain reduced cycling after complete sleep deprivation? Med Sci Sports Exerc. 2013 Dec;45(12):2243-53. doi: 10.1249/MSS.0b013e31829ce379. PMID 23760468
- [Derived] Rabat A, Arnal PJ, Monnard H, Erblang M, Van Beers P, Bougard C, Drogou C, Guillard M, Sauvet F, Leger D, Gomez-Merino D, Chennaoui M. Limited Benefit of Sleep Extension on Cognitive Deficits During Total Sleep Deprivation: Illustration With Two Executive Processes. Front Neurosci. 2019 Jun 19;13:591. doi: 10.3389/fnins.2019.00591. eCollection 2019. PMID 31275098